CLINICAL TRIAL: NCT00234923
Title: A Pilot, Open-Label, Randomized, Comparative Study of the Antiviral Efficacy of Lopinavir/Ritonavir Single-Drug Regimen Versus Lopinavir/Ritonavir in Combination With Lamivudine/Zidovudine in Antiretroviral Naïve Patients
Brief Title: Efficacy and Safety of Kaletra Monotheraphy Compared to Kaletra Based Triple Therapy to Treat HIV in Antiretroviral Naїve Patients
Acronym: MONARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Gerard Goldfarb, Abbott France Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FRAN-03-001; EUDRACT: 2004-816-24; MONARK
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infection
Keywords: HIV Infection; Kaletra; Lopinavir; Ritonavir; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Kaletra Monotherapy: lopinavir/ritonavir
  Interventions: Drug: lopinavir/ritonavir
- 2 (Active Comparator): Kaletra based triple therapy: lopinavir/ritonavir + lamivudine/zidovudine
  Interventions: Drug: lopinavir/ritonavir; Drug: lamivudine/zidovudine

INTERVENTIONS:
Drug: lopinavir/ritonavir — 400 mg lopinavir/ 100 mg ritonavir, BID
  Other Names: ABT-378; Kaletra
Drug: lamivudine/zidovudine — 300mg lamivudine/150mg zidovudine, BID
  Arms: 2

SUMMARY:
The purpose of this pilot study is to obtain a preliminary assessment of the antiviral activity and tolerability of Kaletra single agent therapy as initial treatment for HIV infection, relative to a Kaletra three drug standard of care reference arm

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral naïve
* HIV RNA <100,000 copies/mL
* CD4 cell count >100 cells/mL at screening
* with Karnofsky Score > 70
* If female,

  * non-pregnant and
  * not breastfeeding
* No AIDS opportunistic infection within 30 days of screening

Exclusion Criteria:

* Subject with an HIV primo-infection status
* Recent history of drug and/or alcohol abuse
* History of psychiatric illness
* If presence of the following mutations :

  * in the protease : one among 32,47,48,50,82,84,90
  * OR more than 3 mutations from the other points of the LPV mutation score:10,20,24,46,53,54,63,71
  * in the reverse transcriptase : 215 or 184.
* If abnormal laboratory results such as :

  * Hb<8 g/dl
  * Absolute neutrophil count<750 cells/µl
  * Platelet count<50 000/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2003-08; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Antiviral efficacy by HIV RNA | 48 Weeks

SECONDARY OUTCOMES:
Arm comparisons: CD4 evolution, occurrence of HIV protease and RT mutation, occurrence of AIDS clinical events, safety of NRTI-sparing vs. a PI with 2 NRTIs regimen: clinical and biological tolerance, patient's adherence and quality of life. | 48 weeks
To assess in the LPV/r single-drug regimen arm: virological control, CD4 evolution, safety | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott

REFERENCES:
- [Derived] Tran TA, Ghosn J, Avettand-Fenoel V, Hendel-Chavez H, de Goer de Herve MG, Cohen-Codar I, Rouzioux C, Delfraissy JF, Taoufik Y. Residual HIV-1 replication may impact immune recovery in patients on first-line lopinavir/ritonavir monotherapy. J Antimicrob Chemother. 2015 Sep;70(9):2627-31. doi: 10.1093/jac/dkv138. Epub 2015 May 28. PMID 26023212
- [Derived] Ghosn J, Flandre P, Cohen-Codar I, Girard PM, Chaix ML, Raffi F, Dellamonica P, Ngovan P, Norton M, Delfraissy JF; MONARK Study Group. Long-term (96-week) follow-up of antiretroviral-naive HIV-infected patients treated with first-line lopinavir/ritonavir monotherapy in the MONARK trial. HIV Med. 2010 Feb;11(2):137-42. doi: 10.1111/j.1468-1293.2009.00752.x. Epub 2009 Aug 13. PMID 19682100